CLINICAL TRIAL: NCT01592474
Title: Evolution of Gray Matter Atrophy Over 4 Years in Observational Study of Early IFNβ-1a I.M. Treatment in High Risk Subjects After Clinically Isolated Syndrome (SET Substudy)
Brief Title: Evaluation of Brain Atrophy in CIS Patients on Avonex
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: Biogen (Industry); Jacobs Neurological Institute (Other); Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director, Buffalo Neuroimaging Analysis Center, Professor, University at Buffalo
Other Study IDs: SET
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Avonex; Brain atrophy; MRI; Interferon-beta 1a; IFN Beta 1-a; Clinically isolated syndrome; CIS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is

* To examine if Avaonex can delay the development of clinically definite multiple sclerosis.
* To investigate if Avonex can delay disability progression by slowing brain atrophy.

DETAILED DESCRIPTION:
* Multiple sclerosis (MS) is a chronic inflammatory disorder characterized by focal areas of demyelination in the central nervous system (CNS). MRI findings suggest that we should look at gray matter atrophy as a marker of the disease process in MS.
* Avonex is a proven effective disease-modifying treatment, which reduces total brain and GM atrophy and should be considered first-line therapy in patients with RRMS and CIS.
* The original SET study is an open-label observational study of high risk subjects after CIS for development of CDMS that will enroll 220 patients who have started Avonex immediately after their first clinical attack in Czech Republic, and are followed with clinical and MRI examinations for 4 years at 0, 6, 12, 24, 36 and 48 months. The clinical and MRI acquisition examinations of this study are conducted in Czech Republic.

ELIGIBILITY:
Inclusion Criteria:

* MRI findings must reveal at least 2 hyperintense lesions on T2-WI or FLAIR images at first clinical onset
* CSF examination should confirm oligoclonal bands (examination must be done in an internationally approved lab and the CSF taken before the treatment of attack starts)
* Age 18 - 55 years
* Effective contraception in female patients of childbearing potential
* Kurtzke EDSS ≤ 3.5 at baseline
* Willingness to accept the plan of the study and compliance with the study
* Time from the beginning of first symptoms of CIS to baseline visit should not exceed 4 months (baseline MRI and baseline visit will be organized first 28 days after last steroid administration)
* CIS attack is treated by at least 3g of methylprednisolone without taper
* In case of severe attack 1 g of cyclophosphamide does not disqualify the patient from the study if first MRI and CSF examination was done before treatment administered
* No active major organ disease especially of hepatic or thyroid origin

Exclusion Criteria:

* The clinical diagnosis of MS is definite (the second attack occurs before the baseline visit)
* Age less than 18 or more than 55
* Non-effective contraception method or pregnancy planning
* Active major organ disease, especially hepatic or endocrinologic
* Cooperation of the subject cannot be ensured
* Kurtzke EDSS higher than 3.5 at baseline

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Multiple sclerosis patients being treated with Avonex after first clinical attack.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2005-10; Primary Completion 2011-08 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Can Avonex delay development of clinically definite MS? | 5
  To examine whether Avonex can delay the development of clinically definite multiple sclerosis

SECONDARY OUTCOMES:
Can Avonex delay disability progression? | 5
  To investigate if Avonex can delay disability progression by slowing brain atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD,PhD,FAAN, Principal Investigator — University at Buffalo

REFERENCES:
- [Derived] Ravano V, Andelova M, Fartaria MJ, Mahdi MFA, Marechal B, Meuli R, Uher T, Krasensky J, Vaneckova M, Horakova D, Kober T, Richiardi J. Validating atlas-based lesion disconnectomics in multiple sclerosis: A retrospective multi-centric study. Neuroimage Clin. 2021;32:102817. doi: 10.1016/j.nicl.2021.102817. Epub 2021 Sep 2. PMID 34500427